CLINICAL TRIAL: NCT02103465
Title: Late Onset Parkinson's Disease in Subjects 70 Years and Older: Possible Use of Rotigotine
Brief Title: Possible Use of Rotigotine in Subjects 70 Years and Older With Late Onset of Disease
Acronym: PARROT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Because the rate of recruitment was very slow
Sponsor: Azienda Ospedaliera Cardinale G. Panico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EudraCT Number: 2013-000827-15
Record Dates: First submitted 2014-03-26; First posted 2014-04-04 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; treatment; old patients; Rotigotine
MeSH Terms: conditions — Parkinson Disease | interventions — rotigotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rotigotine (Experimental): 80 patients with late onset PD are randomized in 2 parallel groups, ratio 1:1.
  Interventions: Drug: Rotigotine
- Placebo (Placebo Comparator): 80 patients with late onset PD are randomized in 2 parallel groups, ratio 1:1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rotigotine — transdermal patch
  Other Names: Neupro
  Arms: Rotigotine
Drug: Placebo — transdermal patch
  Arms: Placebo

SUMMARY:
This exploratory trial will fulfill a medical data gap for the dopamine-agonist rotigotine, as so far no data on elderly population is available.

Primary objective: To assess efficacy and safety of rotigotine in patients with late onset Parkinson's Disease (PD), starting at age 70 or later, on motor symptoms.

Secondary objective: To assess efficacy and safety of rotigotine in patients with late onset Parkinson's Disease (PD), starting at age 70 or later, on selected non motor symptoms : sleep quality; depression; cognitive function.

Subjects ≥70 years, with diagnosis of Parkinson's Disease (PD) based on the presence of at least two of three cardinal features (bradykinesia, resting tremor, rigidity), within 12 months since diagnosis and no longer than 12 months from onset to diagnosis, and for whom the caring physician is uncertain on whether or not to start treatment.

Outcome Measurement: Percentage of Responders to treatment in motor (part III) and Activities of daily living (ADL) (part II) components of Unified Parkinson's Disease Rating Scale (UPDRS) at visit 4 and 6; Percentage of Responders to treatment in sleep quality in relation to Parkinson's Disease Sleep Scale (PDSS)-2 at visit 4 and 6; Responders to treatment in mood in relation to Geriatric Depression Scale (GDS) at visit 4 and 6.

Exploratory, randomized, double blind, placebo-controlled study: 80 patients with late onset Parkinson's Disease (PD) are randomized in 2 parallel groups, ratio 1:1.

One group will be treated with rotigotine and one group will be treated with placebo, for 12 weeks after titration.

DETAILED DESCRIPTION:
Treatment is titrated to optimal dose (that at which investigator and subject felt that motor and non motor impairment are adequately controlled), starting at 2 mg/24 hr and increasing with weekly increments of 2 mg/24 hr up to a maximum of 8 mg/24 hr. The dose is maintained at the optimal or maximal dose for a 8-week period (maintenance period) .

ELIGIBILITY:
Inclusion Criteria:

* Age ≥70 years
* Idiopathic Parkinson's Disease (PD) confirmed by at least two of the following signs: resting tremor, bradykinesia, rigidity
* Diagnosis of Parkinson's Disease (PD) within the last 12 months and onset of symptoms within 12 months from diagnosis
* Disease stage I or II according to Hoehn and Yahr Scale
* Ability to provide written informed consent
* Patients willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures

Exclusion Criteria:

* Disease duration more than 12 months since diagnosis and/or duration of symptoms at diagnosis for more than 12 months
* Hoehn & Yahr stage ≥3
* Atypical or secondary parkinsonism
* Patient currently on L-dopa, Dopamine Agonist (DA) or other Parkinson's Disease (PD) medication at baseline
* Centrally acting dopaminergic agents, monoamine oxidase inhibitors (MAOIs), tolcapone, budipine, neuroleptics taken within the 28 days preceding the baseline visit
* History of deep brain stimulation
* History of severe cardiac disease/heart failure in the last 3 years
* History of repeated falls
* History of sulfite sensitivity
* Arterial hypotension
* Stroke or a transient ischemic attack within the last 12 months
* Previous or current treatment with rotigotine (at any time)
* Diagnosis of dementia according to Diagnostic and Statistic Manual (DSM)-IV-Revised
* Mini Mental State Examination (MMSE) total score <24 at screening visit
* History of psychosis
* Clinically relevant hepatic dysfunction and/or transaminase levels 5+ times higher than upper normal value
* Experimental treatments within the antecedent 3 months
* History of drug or alcohol dependency
* Poor compliance with treatment
* Inability to comply with protocol

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Percentage of Responders to treatment (*) in motor (part III) and Activities of daily living (ADL) (part II) components of Unified Parkinson's Disease Rating Scale (UPDRS) at visit 4 and 6 | M2
  (*) Responder to treatment is a subject who has at least a 20% decrease in the sum of scores (parts II and III) from the Unified Parkinson's Disease Rating Scale (UPDRS) subtotal from baseline to the end of the maintenance phase in the direction of normality.
  The outcome will be valuate on Month 2 and Month 4

SECONDARY OUTCOMES:
Percentage of Responders to treatment in sleep quality in relation to Parkinson's Disease Sleep Scale-2 (PDSS) at visit 4 and 6 | M2
  (*) Responder to treatment is a subject who has at least a 20% decrease in the sum of scores (parts II and III) from the Unified Parkinson's Disease Rating Scale (UPDRS) subtotal from baseline to the end of the maintenance phase in the direction of normality The outcome will be valuate on Month 2 and Month 4

OTHER OUTCOMES:
Responders to treatment in mood in relation to Geriatric Depression Scale (GDS) at visit 4 and 6 | M2
  (*) Responder to treatment is a subject who has at least a 20% decrease in the sum of scores (parts II and III) from the Unified Parkinson's Disease Rating Scale (UPDRS) subtotal from baseline to the end of the maintenance phase in the direction of normality.
  The outcome will be valuate on Month 2 and Month 4

CONTACTS AND LOCATIONS:
Overall Officials: Giancarlo Logroscino, Prof, Study Chair — A.O. Ospedale "Card G. Panico" di Tricase
Locations (11):
- Italy (11):
  - Ospedale Lorenzo Bonomo Andria, Andria, Andria-Barletta-Trani
  - Ospedale Generale Regionale "F. Miulli", Acquaviva delle Fonti, Bari
  - Azienda Ospedaliera Universitaria Consorziale Policlinico di Bari, Bari, Bari
  - Ospedale S. Giacomo, Monopoli, Bari
  - Ospedale "A. Perrino", Brindisi, Brindisi
  - A.O. Universitaria "Ospedali Riuniti" - U.O. Neurologia Ospedaliera, Foggia, Foggia
  - A.O. Universitaria "Ospedali Riuniti"-U.O. Neurologia Universitaria, Foggia, Foggia
  - IRCCS "Casa Sollievo della Sofferenza", San Giovanni Rotondo, Foggia
  - Ospedale Francesco Ferrari, Casarano, Lecce
  - Presidio Ospedaliero "Vito Fazzi", Lecce, Lecce
  - A.O. Ospedale "Card. G. Panico" di Tricase, Tricase, Lecce

IPD SHARING:
Plan to Share IPD: No